CLINICAL TRIAL: NCT02386306
Title: A Randomized, Double-Blind, Placebo-Controlled; Phase 1b, Safety, Tolerability, and Pharmacokinetic Study of Multiple Ascending Doses of GC021109 in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Study Evaluating Safety, Tolerability, and PK of Multiple Ascending Doses of GC021109 in Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GliaCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: GC-100-02
Record Dates: First submitted 2015-02-16; First posted 2015-03-11 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2015-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Treatment Cohort 1 (Experimental): Each study participant will be administered with one 1mg dose capsule per day of GC021109 for 28 days.
  Interventions: Drug: GC021109
- Placebo Cohort 1 (Placebo Comparator): Patients receiving placebo as part of each cohort will be dosed with a comparable capsule to those in the treatment arm of each cohort.
  Interventions: Other: Placebo
- Treatment Cohort 2 (Experimental): Each study participant will be administered with one dose per day of GC021109 for 28 days. Dose levels will be determined following a review of cohort 1 safety data through day 14
  Interventions: Drug: GC021109
- Placebo Cohort 2 (Placebo Comparator): Patients receiving placebo as part of each cohort will be dosed with a comparable capsule to those in the treatment arm of each cohort.
  Interventions: Other: Placebo
- Treatment Cohort 3 (Experimental): Each study participant will be administered with one dose per day of GC021109 for 28 days. Dose levels will be determined following a review of cohort 2 safety data through day 14
  Interventions: Drug: GC021109
- Placebo Cohort 3 (Placebo Comparator): Patients receiving placebo as part of each cohort will be dosed with a comparable capsule to those in the treatment arm of each cohort.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GC021109
  Arms: Treatment Cohort 1; Treatment Cohort 2; Treatment Cohort 3
Other: Placebo
  Arms: Placebo Cohort 1; Placebo Cohort 2; Placebo Cohort 3

SUMMARY:
This is a Phase 1b, multi-center, randomized, double-blind, placebo-controlled study designed to evaluate the safety, tolerability, and pharmacokinetics of GC021109 in subjects with mild to moderate Alzheimer's Disease (as determined by 2011 National Institute on Aging- Alzheimer's Association [NIA-AA] criteria and Mini Mental State Examination [MMSE]). The Investigator, study site staff, (with exception of a designated pharmacist/pharmacy technician) and all study subjects will be blinded to randomized study medication assignment until database lock. Treatment assignments may be unblinded for select pre-authorized individuals involved in the safety and PK data reviews in order to accurately determine how to proceed with dose escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 55-85 years, inclusive, at the time of informed consent.
2. Subjects diagnosed with mild to moderate AD as determined by the following:

   1. Diagnosis of probable AD according to the 2011 NIA-AA criteria
   2. MMSE (using serial 7's) score of 12-26 at screening (Mild defined as 20-26 and Moderate defined as 12-19)
   3. Documentation in the clinic notes of mild/moderate AD
3. If on AD therapy, stable dose for at least 3 months prior to screening.
4. All male subjects must practice effective contraception during the study. Females of childbearing potential must use a medically accepted form of birth control, unless postmenopausal for > 1 year (as documented by elevated follicle-stimulating hormone [FSH]) or surgically sterile. All females of childbearing potential must have a negative serum pregnancy test (human chorionic gonadotropin beta [hCGβ]) at screening and a negative urine pregnancy test on Day 1 pre-dose.
5. Body mass index (BMI) between 18 and 35 kg/m2, inclusive, at screening.
6. Must have an eligible caregiver (who spends a minimum of 10 hours per week with the subject) who will be available for the duration of the study to serve as the subject's designee. Caregiver must be willing to comply with study procedures.
7. Caregiver must sign a caregiver ICF after the nature and risks of study participation have been fully explained to them.
8. Patients who are capable, according to the Investigator, or patient's legally authorized representative, must sign a patient ICF after the nature and risks of study participation have been fully explained to them.
9. Patients who are capable of providing assent but not capable of signing the ICF, according to the Investigator, should provide assent for study participation.

   1. Patients who sign the ICF are not required to provide a separate assent.
   2. Patients who are not capable of providing assent are still allowed to participate provided the patient's legally authorized representative agrees to participation.

   Investigators must document the reasons for any patient that is unable to provide assent and maintain this documentation with the consent/assent documents.
10. Must be able to comply with all study requirements and restrictions for the duration of the study.
11. Non-smoker and non-tobacco user for a minimum of 3 months prior to screening and for the duration of the study.
12. Ability to swallow capsules.

Exclusion Criteria:

1. MRI findings inconsistent with AD within the previous 12 months. All subjects must have had a MRI within the previous 12 months to be eligible.
2. History or current evidence of any clinically significant cardiac, endocrinologic, hematologic, hepatobiliary, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease, as determined by the Investigator.
3. History of cancer within the past five years (excluding non-melanoma skin cancer).
4. Active suicidal ideation reported on the Columbia - Suicide Severity Rating Scale (C SSRS) at screening.
5. Clinically significant abnormal laboratory test values at screening (as determined by the Investigator), including:

   1. any values for alanine aminotransferase (ALT) or aspartate aminotransferase (AST) that are 1.5 times above the upper limit of the reference range
   2. any values for total or direct bilirubin that are 1.5 times above the upper limit of the reference range
   3. estimated glomerular filtration rate <85ml/min/1.73m2.
6. Subjects with a QTc of ≥450 msec for males and ≥470 msec for females at screening.
7. Participation in another clinical trial or treatment with an investigational agent within 30 days or 5 half-lives, whichever is longer, prior to Day 1.
8. Subjects with a body weight > 120 kg at screening.
9. History of alcohol or drug abuse or dependence within 12 months of screening as determined by the Investigator.
10. Clinically significant infection within 3 months of screening as determined by the Investigator.
11. Any conditions that, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study.
12. Positive urine screen for prohibited drugs (cocaine, cannabinoids, nicotine [urine cotinine is the detection mechanism for nicotine], opiates, barbiturates, amphetamines, and benzodiazepines) or positive alcohol Breathalyzer on Day 1.
13. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCVAb) at screening.
14. Known or suspected hypersensitivity or idiosyncratic reaction to study medication or any components thereof.
15. Has donated blood within 3 months of screening or plans to donate blood within 3 months of study completion.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Assessment of the number and severity of treatment-emergent AEs (TEAEs) following single oral doses of GC021109 and placebo from Day 1 through Day 28 | 28 days

SECONDARY OUTCOMES:
Estimate of the pharmacokinetic (PK) parameters of multiple, escalating dose levels of GC021109: AUC0-t, AUC0-24, AUC0-inf, AUC%extrap, CL/F, Cmax, Tmax, λz, and t1/2. | 28 days
  Change in plasma PK concentrations will be measured pre-dose through Day 28 of the study and PK parameters derived using non-compartmental and/or compartmental methods as appropriate. The following PK parameters of GC021109 will be calculated: AUC0-t, AUC0-24, AUC0-inf, AUC%extrap, CL/F, Cmax, Tmax, λz, and t1/2.
Determine the effect of multiple, escalating dose levels of GC021109 on potential biomarkers of activities. | 28 days
  Plasma and cerebrospinal fluid samples will be collected pre-dose and on Day 28 to analyze biomarkers such as IL-12, amyloid β, and tau.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Collaborative Neuroscience Network, Long Beach, California
  - Quantum laboratories / Memory Disorder Center, Deerfield Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Compass Research, Orlando, Florida